CLINICAL TRIAL: NCT07190612
Title: Efficacy of Propofol Combination With Either Ketamine, Dexmedetomidine or Midazolam for Sedation During Upper Gastrointestinal Endoscopic Procedures: A Prospective, Randomized, Comparative Study
Brief Title: Efficacy of Propofol Combination With Either Ketamine, Dexmedetomidine or Midazolam for Sedation During Upper Gastrointestinal Endoscopic Procedures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MD228/2024
Record Dates: First submitted 2025-07-24; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-09

CONDITIONS: Upper Gastrointestinal Endoscopy; Anesthesia
Keywords: sedation; ketamine; dexmetomidine; propofol; upper endoscopy; anesthesia; midazolam
MeSH Terms: interventions — Dexmedetomidine; Propofol; Midazolam; Ketamine

STUDY DESIGN:
Intervention Model Description: Three study groups: propofol in combination with either: midazolam, dexmetomidazine, or ketamine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Dexmedetomidine (200 µg/2ml vial) + Propofol (1% 20 mls ampoule)
  Interventions: Drug: Dexmedetomidine and propofol
- Group 2 (Experimental): Ketamine (50mg/1ml vial) + Propofol (1% 20 mls ampoule)
  Interventions: Drug: ketamine and propofol
- Group 3 (Experimental): Midazolam (5mg/1ml ampoule) + Propofol (1% 20 mls ampoule)
  Interventions: Drug: Midazolam and propofol

INTERVENTIONS:
Drug: Dexmedetomidine and propofol — Dexmedetomidine infusion syringe (50mls): will be filled with 2mls of dexmedetomidine (200µg) diluted in 48 ml of 0.9% normal saline to make a final volume of 50mls and a final dexmedetomidine concentration of 4µg/ml. It will be infused as 1µg
  /kg/hr iv. Propofol infusion syringe (50mls): will be filled with 20mls of 1% propofol (200mg) diluted in 30mls 0.9% normal saline to make a final volume of 50mls and a final propofol concentration of 4mg/ml. It will be iv administered as 0.5 mg/kg slow iv for 10 minutes, then infused at a rate of 0.5mg/kg/hr.
  Other Names: Precedex; Diprivan
  Arms: Group 1
Drug: Midazolam and propofol — Midazolam infusion syringe (50mls): will be filled with 10mls of Midazolam (50mg) diluted in 40mls 0.9% normal saline to make a final volume of 50mls to reach a final midazolam concentration of 1mg/ml. It will be administered as a bolus dose of 0.05 mg/kg iv over 2 minutes then infused at a rate of 0.025mg/kg/hr. Propofol infusion syringe (50mls): will be filled with 20mls of 1% propofol (200mg) diluted in 30mls 0.9% normal saline to make a final volume of 50mls and a final propofol concentration of 4mg/ml. It will be iv administered as 0.5 mg/kg slow iv for 10 minutes, then infused at a rate of 0.5mg/kg/hr.
  Other Names: Dormicum; Diprivan
  Arms: Group 3
Drug: ketamine and propofol — Ketamine infusion syringe (50mls): will be filled with 2mls of ketamine (100mg) diluted in 48mls 0.9% normal saline to make a final volume of 50mls to reach a final ketamine concentration of 2mg/ml. It will be administered as a bolus dose of 0.25 mg/kg iv then infused at a rate of 0.25mg/kg/hr. Propofol infusion syringe (50mls): will be filled with 20mls of 1% propofol (200mg) diluted in 30mls 0.9% normal saline to make a final volume of 50mls and a final propofol concentration of 4mg/ml. It will be iv administered as 0.5 mg/kg slow iv for 10 minutes, then infused at a rate of 0.5mg/kg/hr.
  Other Names: Ketam
  Arms: Group 2

SUMMARY:
The investigators are comparing the efficacy of three different sedative agents in gastrointestinal endoscopic procedures.

DETAILED DESCRIPTION:
The investigators aim to compare the efficacy of ketamine-propofol, dexmedetomidine-propofol, and midazolam-propofol combinations as procedural sedative agents for adult patients undergoing elective upper gastrointestinal endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients aged between 18 and 65 years
* Patients who are scheduled for elective upper gastrointestinal endoscopic procedures with sedation
* Patients who are classified as ASA (American Society of Anesthesiologists) I and II

Exclusion Criteria:

* Patient's refusal to participate
* Respiratory compromise as patients with respiratory failure or with active chest conditions, e.g., bronchial asthma or pneumonia
* Cardiovascular compromise including heart failure and shocked patients
* Severe uncontrolled hematemesis with shock or risk of aspiration.
* Patients who are allergic or have any contraindications to any of the used drugs.
* Patients who have a chronic neuropsychiatric disorder or are on a neuropsychiatric drug.
* Patients on long-term sedative medication have a history of drug or alcohol abuse.
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recovery time | From end of drug infusion until recovery (defined as modified Aldrete score ≥9), assessed up to 24 hours postoperatively.
  The time from the stoppage of the drug infusions till achieving a score of≥9 according to the modified Aldrete score.
Induction time | Preoperatively - before the surgery
  The time to reach a sedation level of ≥ 4 on Ramsay's sedation score.

SECONDARY OUTCOMES:
Mean arterial pressure (MAP)(mmHg) | perioperatively
  systolic blood pressure (SBP) (mmHg) and diastolic blood pressure (DBP) (mmHg) recorded to calculate the Mean arterial pressure
Ramsay Sedation Scale | Every 5 minutes from the start of the procedure until its completion, assessed up to 4 hours.
  All patients will be targeted to reach deep sedation defined as a Ramsay Sedation Scale score of ≥4 (scale range: 1-6; 1 = anxious/awake, 6 = no response to stimuli).
Endoscopist satisfaction | Perioperatively
  Endoscopist assessment of the sedation as excellent/good/not bad/bad
Endoscopy procedure time | Peri- operatively
  The duration of time the endoscope was in the oral orifice.
Rescue propofol total doses (mg) | Perioperatively
  In the case of RSS<4 or if the patient shows limb movement at any time within the procedure, propofol 20 mg IV increments will be given, and total given doses in mg will be recorded
Sedation-related adverse effects (SRAEs) and complications | Perioperatively
  Any incidence of respiratory (e.g. apnea, desaturation) or hemodynamic compromise (e.g hypotension, bradycardia, tachycardia, arrhythmia, cardiac arrest) or any other adverse effects (e.g. nausea, vomiting, allergy, seizure, recovery agitation, and delayed recovery) will be managed accordingly and documented.
Heart rate | Perioperatively
  (beats/min)
Peripheral oxygen saturation (SPO2) | Perioperatively
  oxygen %

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Mohammad, Msc., Principal Investigator — AinShams University

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality

DOCUMENTS (3):
  • Study Protocol (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT07190612/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT07190612/SAP_001.pdf
  • Informed Consent Form (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT07190612/ICF_002.pdf